

# **DEPARTMENT OF HEALTH & HUMAN SERVICES**

Public Health Service

National Institutes of Health Bethesda, Maryland 20892

www.nih.gov

Date: 5/24/2024

To: The A5332 Protocol Team, Principal Investigators and Study Coordinators

Jui Shah, Ph.D., Chief Protection of Participants, Evaluation, and Policy

From: Branch (ProPEP), Division of AIDS

A5332, Version 6.0 – Final – Spanish Sample Informed Consent dated 16 May

Subject: 2022

The purpose of this letter from the **Protection of Participants, Evaluation, and Policy Branch** of the Division of AIDS is to document that the Spanish Sample Informed Consent provided in protocol A5332, Version 6.0 is a complete and accurate translation of the English Sample Informed Consent. The Spanish Sample Informed Consent contains all the required Basic and Additional elements of an Informed Consent required by the Code of Federal Regulations.

The translation of the English Sample Informed Consent into Spanish was performed by one of the qualified English to Spanish Translators supported by the DAIDS Regulatory Support Contract (RSC). The English to Spanish Translators have excellent qualifications and have passed a quality assurance translation test facilitated by the NIH Translation Unit.

## Consent Forms:

- Appendix I: Sample Informed Consent
- Appendix IA: Sampled Informed Consent Addendum

## APÉNDICE I: MODELO DE CONSENTIMIENTO INFORMADO

Para el Protocolo REPRIEVE (A5332), Versión FINAL 6.0, del 16 de mayo de 202

Ensayo Clínico Aleatorizado para Prevenir Eventos Vasculares en el VIH (El Estudio REPRIEVE)

## INTRODUCCIÓN

Se le solicita a usted que participe en este estudio de investigación debido a que usted **vive** con el virus de la inmunodeficiencia humana (VIH), el virus que causa el SIDA, y está tomando medicamentos contra el VIH.

Este estudio es patrocinado por los Institutos Nacionales de la Salud (NIH, siglas en inglés). El/La médico(a) a cargo de este estudio en este sitio es: (inserte el nombre del Investigador Principal). Antes de que usted decida si quiere ser parte de este estudio, nosotros queremos que sepa en qué consiste el estudio.

## ¿PARA QUÉ SE LLEVA A CABO ESTE ESTUDIO?

Desde que las personas comenzaron a tomar medicamentos contra el VIH, las enfermedades causadas por el SIDA han disminuido, pero otras enfermedades graves, como la enfermedad cardiaca, han aumentado. El VIH causa inflamación (irritación) dentro del organismo, que no puede sentirse pero se puede medir. Estas pruebas se describirán más adelante en este formulario de consentimiento. La inflamación puede contribuir a desarrollar dolencias tales como la enfermedad cardiaca, que se ha vuelto una de las causas principales de muerte en personas con VIH (PWH, siglas en inglés). Los medicamentos contra el VIH pueden reducir la inflamación de cierta manera, sin embargo a veces los niveles de inflamación pueden permanecer altos si se comparan con el de personas sin el VIH.

Las estatinas son un grupo de medicamentos que se utilizan para reducir los niveles de colesterol y triglicéridos (grasas en la sangre) que generan las personas, y para prevenir eventos relacionados con las enfermedades del corazón, tales como ataques cardiacos, en el caso de personas que tienen un alto riesgo de sufrir ataques cardiacos. Los estudios han demostrado que las estatinas pueden tener otros beneficios; por ejemplo, disminuyendo los niveles de inflamación, las estatinas pueden tener un efecto protector contra las enfermedades cardiacas y los eventos relacionados con éstas. Asimismo, las estatinas pueden tener algunos efectos beneficiosos en algunas otras enfermedades como ciertos tipos de cáncer o problemas renales.

Las pautas más recientes del Colegio Americano de Cardiología y la Asociación Americana del Corazón (ACC/AHA, siglas en inglés) recomiendan el uso de estatinas si alguien está en riesgo de sufrir una enfermedad relacionada con el corazón, en base a varios factores diferentes, incluyendo el uso de una calculadora de riesgos basada en factores de riesgo conocidos como sexo, edad, raza, niveles de colesterol, consumo de tabaco, diabetes e hipertensión, que estima el riesgo a 10 años de sufrir ataque cardiaco, apoplejía u otro evento (la puntuación de riesgo

ASCVD, siglas en inglés). La infección por VIH no está incluida en la calculadora de riesgo. Las actuales calculadoras de riesgo no pueden predecir con precisión el riesgo en las **PWH**. Sin embargo, la infección por VIH, los medicamentos contra el VIH y la inflamación crónica pueden poner a usted en un riesgo más alto de sufrir estas enfermedades, aunque no sabemos si usted se beneficiaría al tomar estatinas. Usted es elegible para este estudio porque está en el grupo de riesgo bajo a moderado de sufrir enfermedad cardiaca, según las pautas actuales, y no existe consenso respecto a que las **PWH** en este grupo debieran tomar estatinas. Su participación en este estudio nos ayudará a determinar si el uso de las estatinas puede prevenir enfermedades relacionadas con el corazón entre las **PWH**. Los resultados de este estudio pueden ayudar a crear pautas de prevención de la enfermedad cardiaca en la infección por VIH.

Para las personas VIH negativas con una puntuación de riesgo ASCVD de entre 7,5% y 15%, las pautas actuales recomiendan una discusión entre el proveedor de salud y los pacientes sobre los riesgos y beneficios de la terapia con estatinas y aconsejan iniciar las estatinas sobre la base de los datos de los ensayos clínicos disponibles. Sin embargo, para las **PWH** y un riesgo moderado de enfermedad cardiaca (una puntuación de riesgo entre 7,5% y 15%), no hay actualmente datos disponibles que nos digan con claridad si los beneficios de la terapia con estatinas superan a los riesgos, incluidos los efectos secundarios y las potenciales interacciones de medicamento a medicamento. Algunos proveedores de salud pueden elegir la terapia con estatinas para el tratamiento de **PWH** en este rango de riesgo moderado, y esta opción puede estar disponible para usted, en lugar de participar en el ensayo clínico. En última instancia, los resultados de este ensayo proporcionarán datos para guiar el uso de estatinas en las **PWH**.

La pitavastatina es una estatina que, junto a una dieta, ha sido aprobada por la Administración de Alimentos y Medicamentos de los Estados Unidos para tratar el colesterol alto. También disminuye los niveles de triglicéridos en la sangre. No ha sido estudiada para ver si reduce las enfermedades relacionadas con el corazón o la mortalidad. Se eligió la pitavastatina porque se estima que hay pocas interacciones entre la pitavastatina y los medicamentos que se usan habitualmente para tratar el VIH.

El propósito principal de este ensayo clínico es observar si la pitavastatina puede prevenir la enfermedad cardiaca y las muertes por causas cardiacas en **PWH** que están tomando medicamentos contra el VIH. También evaluaremos la seguridad de la pitavastatina.

¿CUÁNTAS PERSONAS ESTARÁN EN ESTE ESTUDIO?

Alrededor de 7500 personas participarán en este estudio.

¿QUÉ DEBO HACER SI ESTOY EN ESTE ESTUDIO?

#### Visitas del estudio

Si usted ingresa al estudio, será observado(a) en la clínica alrededor de 6 veces durante el primer año. Posteriormente, las visitas del estudio serán cada 4 meses durante los siguientes 6 a 10 años, según cuándo se incorpore. El personal del estudio le informará cuánto tiempo

durará cada visita. Más detalles sobre las visitas y procedimientos del estudio se le brindan a continuación.

## Si usted no ingresa en el estudio

Si usted decide no participar en este estudio después de firmar el formulario de consentimiento, o si usted no cumple con los requisitos de elegibilidad, nosotros usaremos parte de la información sobre usted. Como parte de esta visita de tamizaje, se obtiene de usted cierta información demográfica (por ejemplo, edad, sexo, raza), clínica (por ejemplo, condición de la enfermedad, diagnóstico) y de laboratorio (por ejemplo, análisis de seguridad), de modo que los investigadores del Grupo de Ensayos Clínicos de SIDA (ACTG, siglas en inglés) puedan ayudar a determinar si hay patrones o razones comunes por las cuales las personas no se incorporan a un estudio.

## Medicamentos del estudio

Si usted ingresa al estudio, será asignado(a) aleatoriamente (como al lanzar una moneda al aire) para recibir ya sea la pitavastatina o el placebo de pitavastatina. El placebo es un comprimido que se parece a la pitavastatina pero no contiene en él ningún medicamento activo. Por lo tanto, existe la probabilidad de que si usted es aleatorizado(a) para tomar el placebo no reciba el tratamiento durante su participación en el estudio. En los ensayos clínicos usamos placebos para saber si los efectos que se observan en el ensayo se deben realmente al medicamento del estudio o a otras razones. Ni usted ni el personal del estudio conocerán su asignación. Usted no conocerá su asignación hasta después de que todo el estudio finalice y los resultados del estudio se den a conocer. En el caso de que sea necesario para su salud, se le dará a conocer a usted y su médico(a) su asignación.

Usted tomará el medicamento del estudio (ya sea la pitavastatina o el placebo de pitavastatina) una vez al día, todos los días, durante el período del estudio, con o sin comida. La dosis es de 4 mg. Le recomendamos que tome el medicamento del estudio cada día a la misma hora. El estudio suministra estos medicamentos. Es muy importante que usted tome los medicamentos como se le indicó. En cada visita del estudio posterior al ingreso, le preguntaremos cómo ha estado tomando sus medicamentos del estudio. Los medicamentos antirretrovirales (tratamiento del VIH) no serán suministrados por el estudio.

#### Procedimientos del estudio

El personal del estudio puede contestar cualquier pregunta que usted tenga acerca de las visitas de estudio individuales y los procedimientos. La tabla siguiente se puede utilizar como una referencia rápida, junto con las explicaciones que siguen.

Apéndice I, Tabla 1: Procedimientos del Estudio

| Procedimiento | Tamizaje¹ | Ingreso <sup>2</sup> | Mes 1 | Visitas cada 4<br>meses (inician<br>en el mes 4) | Visitas<br>anuales<br>(inician en<br>el mes 12) | Visita final |
|---|---|---|---|---|---|---|
| Examen físico | X | | X | | Х | Х |
| Evaluación de riesgo de enfermedad cardiaca | Х | | | | | |
| Factores de riesgo de | Х | | | | | |

| Procedimiento | Tamizaje <sup>1</sup> | Ingreso <sup>2</sup> | Mes 1 | Visitas cada 4<br>meses (inician<br>en el mes 4) | Visitas<br>anuales<br>(inician en<br>el mes 12) | Visita final |
|---|---|---|---|---|---|---|
| enfermedad cardiaca | | | | | | |
| Preguntas sobre dieta y ejercicios | | X | | | | X |
| Información para cambiar el estilo de vida | | X | | | Х | X |
| Preguntas sobre la salud y los medicamentos | X <sup>3</sup> | Х | Х | X <sup>5</sup> | X <sup>5</sup> | X <sup>3,5</sup> |
| Extracción de sangre | X | X | X | | X | X |
| Obtención de orina | | Х | | | X <sup>4</sup> | |
| Análisis de embarazo | Х | Х | Х | Х | Х | Х |
| Electrocardiograma | | Х | | | | |
| Píldoras dispensadas | | х | | Х | Х | |

<sup>&</sup>lt;sup>1</sup> Visita de tamizaje: antes de que usted pueda entrar al estudio, deberá venir a la clínica para que se le hagan evaluaciones y así asegurarnos de que pueda participar del estudio.

Si usted deja el estudio antes de tiempo, o tiene que dejar de tomar el medicamento del estudio antes de que éste finalice, se le harán a usted los procedimientos de la siguiente tabla. Apéndice I, Tabla 2: Discontinuación de los Procedimientos del Estudio

| Procedimiento | Interrupción prematura del estudio o del tratamiento del estudio |
|---|---|
| Examen físico | X |
| Preguntas sobre salud y medicamentos | X <sup>1</sup> |
| Análisis de embarazo | X |
| Extracción de sangre | X |
| Análisis de sangre en ayunas | X |

Esto también incluirá una evaluación hormonal de las mujeres y una evaluación de COVID-19 en todos los participantes.

Explicación de los procedimientos del estudio

## Examen físico

<sup>&</sup>lt;sup>1</sup> Visita de ingreso: si usted cumple con los requisitos para el ingreso, usted se inscribirá en el estudio.

<sup>&</sup>lt;sup>2</sup> Esto incluirá también una evaluación hormonal de las mujeres.

<sup>&</sup>lt;sup>3</sup> SOLO sitios del ACTG: se obtendrá orina en los meses 12, 24 y 48 solo de las personas inscriptas en REPRIEVE (A5332) antes del 1 de enero de 2018.

<sup>&</sup>lt;sup>4</sup> Esto incluirá también una evaluación de COVID-19 en todos los participantes.

Se le realizará a usted un examen físico en el tamizaje. En otras visitas posteriores al ingreso, la extensión del examen dependerá de cómo se sienta en esa visita. Se le controlarán los signos vitales, incluyendo la presión sanguínea y el pulso. Se le medirá su cintura, peso y estatura. Se le preguntará sobre su salud y sus medicamentos.

## Evaluación del riesgo de enfermedad cardiaca

En el tamizaje, le haremos preguntas específicas para evaluar la elegibilidad en base al riesgo de que sufra una enfermedad cardiovascular. En el tamizaje, a usted también se le harán preguntas sobre factores de riesgo cardiovascular, incluyendo sus antecedentes familiares, si fuma, bebe alcohol, consume drogas, dieta y ejercicio.

#### Estilo de vida /orientación y apoyo psicológico para reducir el riesgo

Si usted se incorpora al estudio, se le dará información sobre una dieta sana y la importancia de hacer ejercicio, dejar de fumar, seguir su terapia antirretroviral y tomar el medicamento del estudio tal como se le indicaron. Le daremos esta información en todas las visitas anuales.

#### **ECG**

En el ingreso, se realizará un electrocardiograma o ECG. Un ECG es un registro de la actividad eléctrica de su corazón, que puede mostrar con qué esfuerzo está funcionando. Usted se acostará sin moverse durante no más de 10 minutos mientras se lleva a cabo el ECG.

#### Extracción de sangre

Se le extraerá sangre para diferentes análisis, si no están disponibles como parte de su atención médica de rutina, o bien por cuestiones de seguridad. Se incluirán análisis de rutina para evaluar recuentos sanguíneos, el hígado y la función renal.

En el tamizaje, usaremos los resultados de sus pruebas de la función hepática efectuadas como parte de su atención de rutina por su proveedor de salud. En el mes 1 y el mes 12, a usted le extraeremos sangre para evaluar su función hepática. Este análisis se exige como parte de su participación en el estudio. En cada una de estas visitas, se le extraerá aproximadamente 1 cucharadita de sangre para efectuar este análisis.

En el tamizaje y en la visita final del estudio usaremos los resultados de su CBC (siglas en inglés de recuento de sangre) y función renal, obtenidos por su proveedor de salud como parte de la atención de rutina.

En el tamizaje y en las visitas anuales, usaremos los resultados de su recuento de linfocitos T CD4 (cuántas células que combaten las infecciones hay en su sangre), obtenidos por su proveedor de salud como parte de la atención de rutina.

En el ingreso y en las visitas anuales usaremos los resultados de la carga viral del VIH (cuánto VIH hay en su sangre), obtenidos por su proveedor de salud como parte de la atención de rutina.

En el tamizaje, usaremos los resultados de los niveles de colesterol (grasas que se hallan en la sangre) realizados por su proveedor de salud como parte de su atención de rutina.

Se le darán a conocer los resultados de estos análisis de rutina.

En el ingreso, en todas las visitas anuales, y en la visita final del estudio, se le extraerá algo de sangre y se la almacenará para análisis que se efectuarán más adelante en el estudio o después de que finalice el estudio. Estos análisis medirán los niveles de grasas y azúcar en la sangre. Algunos de esos análisis se usarán para hacer análisis metabólicos en la sangre (que miden de qué manera su organismo usa la comida que usted ingiere). Usted no tiene la obligación de aceptar que se almacene esta sangre para incorporarse al estudio y puede cambiar de opinión sobre el almacenamiento de la sangre cuando lo desee. Su sangre se puede almacenar (con los protectores usuales de la identidad) por tiempo indefinido. No se le darán a conocer los resultados de la investigación que se realice con su sangre.

En cada una de estas visitas, se le extraerán y almacenarán aproximadamente 2 cucharaditas de sangre con estos propósitos.

| ¿Acepta ust<br>grasas y azı | • | | sus muestras para l | hacer pruebas que midan los nive | les de |
|---|---|---|---|---|---|
| S | í | _NO | Iniciales | | |
| Estudio) y e investigación enfermedad no tiene la custed puede sangre se proposition en la custed puede sangre se proposition de la custed puede sangre se proposition de la custed puede sangre se proposition de la custed puede se proposition de la custe de la custed puede se proposition de la custe | n la visita fi<br>n aprobada<br>es cardiova<br>obligación de<br>cambiar de<br>uede almac | nal del estud<br>por REPRIE<br>sculares, VII<br>e aceptar que<br>e opinión sob<br>enar (con los | io, algo de sangre s<br>VE (siglas en inglés<br>H, inflamación, cánd<br>e se almacene esta<br>pre el almacenamien<br>s protectores usuales | ó en la tabla de Procedimientos de se extraerá y almacenará para futus) sobre distintas afecciones, como cer o medicación con estatinas. Un sangre para incorporarse al estudito de sangre cuando lo desee. Ses de la identidad) por tiempo indeción que se realice con su sangre. | ura<br>Io<br>Jsted<br>dio y<br>Su<br>efinido |
| Hasta <b>15</b> cu<br>propósitos. | charaditas | de sangre se | e obtendrán en <b>cada</b> | a una de estas visitas para estos | ; |
| tales como estatinas? | enfermedad | | sculares, VIH, inflam | futura investigación sobre afeccion<br>nación, cáncer y medicación con | nes |

Todos los sitios de ACTG agregarán a su consentimiento local: Se le extraerá alrededor de 1 cucharadita de sangre para observar los genes que pueden afectar el riesgo de sufrir enfermedad cardiovascular y cómo las estatinas actúan en su organismo. Los análisis genéticos son pruebas de laboratorio que observan las diferencias entre los genes de las personas. Su organismo, como el de todos los seres vivos, está hecho de células, y las células contienen ácido desoxirribonucleico, también conocido como "ADN". El ADN es como una cadena de información reunida en un orden determinado. Las partes de la cadena constituyen "genes". Los genes contienen instrucciones sobre cómo su organismo debe funcionar y combatir las enfermedades. Los análisis en este estudio se enfocarán en ciertos genes que se sabe que tienen un efecto sobre las enfermedades cardiovasculares y de qué manera su

7

organismo usa las estatinas. Es posible que en el futuro se identifiquen nuevos genes de interés y que también puedan ser examinados.

Su conformación genética es solo suya, de modo que existe el riesgo en la investigación genética de que, a pesar de todas las medidas de seguridad que se tomen, alguien que use sus muestras o su información genética pueda averiguar que esa información es de usted. Sin embargo, este riesgo es muy pequeño, aunque se puede incrementar con el tiempo, dado que la ciencia y la tecnología progresan rápidamente.

SOLO los sitios de ACTG en los Estados Unidos agregarán a su consentimiento local: En el caso de que la información genética sobre usted sea vinculada con su nombre, la ley federal de los Estados Unidos denominada Ley de No Discriminación por Información Genética (GINA, siglas en inglés), le ayuda a protegerse. Esta norma prohíbe a las compañías de seguro de salud, a los planes de salud de grupos y a la mayoría de los empleadores, negarse a brindar servicios en base a su información genética. Sin embargo, la ley GINA no le protege a usted contra la discriminación que pueda sufrir por parte de compañías que venden seguros de vida, seguros por discapacidad o seguros de cuidados de largo plazo.

| Todos los sitios de ACTG agregarán esta opción para el participante en su consentimiento local: Nos gustaría utilizar parte de la sangre que obtenemos de usted para observar sus genes (ADN). ¿Usted está de acuerdo con este estudio genético? |
|---|
| SINOIniciales |

Si en una fecha posterior usted cambia de parecer y quiere que se destruyan sus muestras, contacte al personal de la investigación. Hay dos formas de retirar su autorización. Usted podría autorizar a los investigadores a que retiren todos los identificadores personales de sus muestras, de modo que estas no se puedan vincular más con usted. Estas muestras se volverán anónimas. O bien, usted puede pedirles a los investigadores que destruyan sus muestras, de modo que no se puedan usar en futura investigación. Sin embargo, cualquiera sea el caso, los investigadores no podrán destruir las muestras o la información de la investigación que ya se esté llevando a cabo.

Para todos los sitios fuera de los Estados Unidos, agregar a su consentimiento local: Sus muestras se pueden enviar y almacenar fuera de su país y pueden ser usadas por investigadores fuera de su país.

## Obtención de orina

Se obtendrá orina en el ingreso para controlar las proteínas en su orina. Los resultados de este análisis no se conocerán inmediatamente; por lo tanto, no le podemos asegurar que se le darán a conocer los resultados de este análisis.

inscriptos en REPRIEVE (A5332) antes del 1 de enero de 2018, también se recogerá orina en los meses 12, 24 y 48, para controlar su función renal.

#### Análisis de sangre en ayunas

Antes del tamizaje, en el ingreso y en todas las visitas anuales, usted no debe comer ni beber nada, incluida cualquier clase de comida, bebidas, caramelos o goma de mascar, durante 8 horas antes de la visita. Se le aconseja que tome agua antes de sus visitas. Si usted no está en ayunas, le pediremos que regrese en ayunas para que se le extraiga sangre dentro de los 30 días de la visita del estudio.

#### Medicamentos del estudio que se le darán a usted

Los medicamentos del estudio se le darán a usted en el ingreso y cada 4 meses. No se le darán a usted medicamentos del estudio en la visita final del estudio.

#### Cuestionarios

Se le preguntará sobre su dieta y ejercicios en el ingreso y esto se repetirá en la visita final del estudio.

¿POR CUÁNTO TIEMPO ESTARÉ EN ESTE ESTUDIO?

Usted estará en este estudio alrededor de 6 a 10 años (72 a 120 meses) según cuándo se incorpore.

# ¿POR QUÉ PODRÍA EL/LA MÉDICO(A) APARTARME DE ESTE ESTUDIO ANTES DE TIEMPO?

El/La médico(a) del estudio puede necesitar apartarlo(a) del estudio antes de tiempo sin su permiso si:

- El/la médico(a) cree que es lo más conveniente para usted.
- Se cancela el estudio.
- Usted no puede concurrir a las visitas del estudio tal como lo requiere el estudio.

El/La médico(a) del estudio puede necesitar retirarle el medicamento del estudio sin su permiso si:

- Usted no puede tomar el medicamento del estudio tal como lo requiere el estudio.
- Continuar con el medicamento del estudio puede ser perjudicial para usted.
- Usted necesita un tratamiento que no puede recibir mientras esté en el estudio.
- Usted gueda encinta.

Si usted debe dejar de tomar el medicamento del estudio antes de que finalice el estudio, le pediremos que continúe participando del estudio y que regrese para algunas visitas y procedimientos del estudio.

Si usted tiene que dejar de tomar de forma permanente el medicamento del estudio, o una vez que deje el estudio, ¿cómo se le proveerá la pitavastatina?

#### Durante el estudio:

Si usted debe dejar de recibir de forma permanente el medicamento pitavastatina suministrado por el estudio antes de que finalice su participación en el estudio, el personal del estudio analizará otras opciones que puedan beneficiarlo(a). Si usted descontinúa su participación activa en el estudio, el personal del estudio se pondrá en contacto anualmente con usted, sus contactos provistos, el departamento de registros médicos o su proveedor de salud, para determinar si usted ha tenido alguna enfermedad cardíaca, accidente cerebrovascular o enfermedad vascular, o si ha fallecido (y la causa de la muerte desde el último contacto).

## Después del estudio:

Después de que usted haya completado su participación en el estudio, éste no podrá seguir suministrándole a usted la pitavastatina que usted recibía en el estudio. Si continuar tomando éste o similares medicamentos pudiera ser beneficioso para usted, el personal del estudio analizará cómo puede hacer usted para obtenerla. ¿CUÁLES SON LOS RIESGOS DEL ESTUDIO?

El medicamento usado en este estudio puede tener efectos secundarios, algunos de los cuales se enumeran a continuación. Tenga en cuenta que estas listas no incluyen todos los efectos secundarios observados con este medicamento. Estas listas incluyen los efectos secundarios más graves o habituales con una relación conocida o posible. Si usted tiene preguntas respecto a los efectos adicionales del medicamento del estudio, pregúntele al personal médico de su sitio.

Existe el riesgo de sufrir efectos secundarios graves o peligrosos para la vida, cuando medicamentos que no son del estudio se toman junto con el medicamento del estudio. Por su seguridad, usted debe informarle a el/la médico(a) o enfermero(a) del estudio sobre todos los medicamentos que se encuentre tomando antes de comenzar el estudio y además antes de comenzar a tomar cualquier nuevo medicamento mientras esté en el estudio. Asimismo, antes de inscribirse en cualquier otro ensayo clínico, usted debe informárselo a el/la médico(a) o enfermero(a) del estudio mientras se encuentre en este estudio.

#### Riesgos de la Pitavastatina

- Problemas musculares. La pitavastatina ocasionalmente puede causar graves problemas musculares, que pueden ocasionar problemas renales, incluyendo insuficiencia renal y rara vez la muerte.
- Problemas hepáticos. La pitavastatina ocasionalmente puede causar problemas hepáticos, que rara vez pueden ser graves u ocasionar la muerte. Su enfermero(a) o médico(a) del estudio le realizará análisis de sangre para controlar su hígado antes de comenzar a tomar la pitavastatina y mientras usted se encuentre tomándola.
- Asegúrese de informar a su médico(a) o enfermero(a) del estudio de inmediato si usted tiene alguno de los siguientes problemas:
- Problemas musculares, como debilidad, sensibilidad, o dolores que aparecen sin una razón aparente, especialmente si usted también tiene fiebre o siente más cansancio que el habitual.
- Náuseas y vómitos.
- Orina de tonalidad marrón o de color oscuro.
- Sentir más cansancio que el habitual.
- Notar que la piel y la parte blanca de los ojos se tornan amarillas.
- Tener dolor de estómago.

Otros problemas que han sido ocasionados por la pitavastatina son dolores de cabeza, salpullido (que rara vez puede ser grave o fatal), reacción alérgica grave o hinchazón, estreñimiento, gases, diarrea, dolor o entumecimiento en los brazos o las piernas, ruptura de tendón, infección del tracto urinario, mareos, deterioro de la memoria y depresión. Todos estos problemas son de infrecuentes a raros.

#### Riesgos de las extracciones de sangre

Extraer sangre puede causar cierto malestar, vahídos, sangrado, hinchazón o moretones donde la aguja penetra en el cuerpo, y en casos raros, desmayos o infección.

#### Riesgos del ayuno

Algunas personas encuentran que ayunar puede ser muy molesto. Puede hacer que algunos individuos se sientan ansiosos, irritables o hambrientos. Los pacientes a los que se les exigen que tomen sus medicamentos matutinos con comida deberían esperar hasta después de completar la visita para tomar sus medicamentos.

#### Riesgos del ECG

Usted puede sufrir una irritación leve, un enrojecimiento ligero y picazón en la piel donde se colocan los electrodos del electrocardiógrafo.

TODOS los sitios de ACTG agregarán a su consentimiento local:

#### Análisis Genéticos

Los resultados de sus pruebas genéticas son sólo para fines de investigación y los resultados individuales no serán devueltos a usted. Los resultados de los estudios genéticos nunca formaran parte de su historia clínica. Vamos a proteger su confidencialidad en la mayor medida. Las muestras de sangre para estudios genéticos serán identificadas de modo tal de mantener su confidencialidad.

| Los resultados del estudio de investigación no se les darán a miembros de su familia, |
|---|
| compañías de seguro, empleadores, o terceros, sin su permiso por escrito y la aprobación de la |
| Junta Institucional de Revisión en |

## Riesgos desconocidos

Podrían presentarse durante el estudio otros efectos secundarios desconocidos en este momento. Todos los medicamentos tienen un posible riesgo de reacción alérgica, que si no se trata de inmediato podría poner la vida en peligro. Durante el estudio, se le dará a conocer cualquier nueva información que pueda afectar su decisión de permanecer en el estudio. Si usted decide permanecer en el estudio, se le pedirá que firme un formulario de consentimiento actualizado. Si usted decide dejar el estudio antes de tiempo, el personal del estudio hablará con usted sobre sus opciones de tratamiento.

## ¿HAY RIESGOS RELACIONADOS CON EL EMBARAZO?

La pitavastatina es insegura para los bebés en gestación. Los riesgos para los bebés en

gestación incluyen defectos de nacimiento, parto prematuro o la muerte. Si usted mantiene relaciones sexuales que pudieran conducir a un embarazo, usted debe aceptar no quedar encinta.

Si usted puede quedar encinta, usted se debe hacer un análisis de embarazo antes de que ingrese a este estudio y en cada visita (se obtendrá 1 cucharadita de sangre o una muestra de orina) y en cada oportunidad en que se sospeche un embarazo. Este análisis debe indicar que usted no está encinta. Si usted queda encinta o piensa que puede estar encinta en cualquier momento durante el estudio, dígaselo de inmediato al personal del estudio. El personal del estudio hablará con usted sobre sus opciones.

Debido al riesgo involucrado, usted y su pareja deben usar al menos un método aceptado de control de la natalidad que usted analice con el personal del estudio. Usted debe comenzar a usar un método aceptado de control de la natalidad al menos dos semanas antes de que comience a tomar el medicamento del estudio y continuar usando una forma aceptada de control natal hasta al menos 6 semanas después de haber interrumpido el medicamento del estudio. Si usted mantiene relaciones sexuales que puedan causar un embarazo, y no usa ninguna forma aceptada de control natal, su médico(a) del estudio le retirará el medicamento del estudio. Usted puede elegir alguno de los siguientes métodos de control natal que se enumeran a continuación:

- Condones (masculinos o femeninos), con o sin un agente espermicida
- Un diafragma o capuchón cervical, con espermicida
- Un DIU (dispositivo intrauterino)
- Ligadura de trompas
- Microinsertos en las trompas
- Anticoncepción de base hormonal

Si usted queda encinta durante el estudio, el personal del estudio querría obtener información sobre el resultado de su embarazo (incluso si éste es posterior a que deje el estudio). Si usted está tomando medicamentos contra el VIH cuando queda encinta, su embarazo será informado a una base de datos internacional que recopila información sobre embarazos de mujeres que toman medicamentos contra el VIH. Este informe no usará su nombre ni ninguna otra información que pudiera identificarla.

#### Lactancia

Se desconoce si el medicamento del estudio pasa a través de la leche materna y puede causar un daño al lactante. Las mujeres que comienzan a dar de lactar deben dejar de tomar el medicamento que suministra el estudio.

## ¿HAY BENEFICIOS AL PARTICIPAR EN ESTE ESTUDIO?

Los estudios han demostrado que las estatinas brindan un beneficio en términos de prevención de enfermedades cardiacas en **personas sin** el VIH con inflamación, pero los efectos de las estatinas para prevenir enfermedades cardiacas en **PWH** es desconocida. Si usted participa en este estudio, puede haber un beneficio directo para usted, pero no se le pueden brindar garantías. Es posible que usted obtenga un beneficio al conocer su riesgo de sufrir un evento cardiovascular, pero también es posible que usted no reciba ningún beneficio por estar en este

estudio, ya sea porque el medicamento no puede funcionar o porque a usted se le asignó el placebo. La información adquirida en este estudio puede ayudar a otras personas que tienen el VIH y están en riesgo de sufrir enfermedad cardiovascular.

# ¿QUÉ OTRAS OPCIONES TENGO ADEMÁS DE ESTE ESTUDIO?

En lugar de estar en este estudio, usted tiene la opción de:

- Tratamiento con medicamentos recetados disponibles para usted
- Tratamiento con medicamentos experimentales, si usted califica
- Ningún tratamiento
- Continuar con la atención médica de rutina que le brinda su proveedor de atención primaria
- Incorporarse a otro ensayo clínico, si usted califica
- No recibir atención médica

Hable con el/la médico(a) del estudio sobre estas y otras opciones disponibles para usted. Su médico(a) del estudio le explicará los riesgos y beneficios de estas opciones. ¿QUÉ HAY QUE SABER ACERCA DE LA CONFIDENCIALIDAD?

Para TODOS los sitios de los Estados Unidos: Nosotros haremos todo lo posible para proteger su privacidad. Además de los esfuerzos del personal del estudio para ayudar a mantener en reserva su información personal, hemos obtenido un Certificado de Confidencialidad del Gobierno Federal de los Estados Unidos. Este Certificado implica que los investigadores no pueden ser obligados a informarles sobre su participación a personas que no estén conectadas con este estudio, tales como los miembros del sistema judicial. Asimismo, ninguna publicación de este estudio utilizará su nombre ni lo/la identificará a usted personalmente.

Las personas que pueden revisar sus expedientes incluyen al Grupo de Ensayos Clínicos de SIDA (ACTG), la Oficina para la Protección de los Seres Humanos en la Investigación (OHRP, siglas en inglés) u otras agencias gubernamentales como parte de sus obligaciones, la Administración de Alimentos y Medicamentos (FDA), la IRB (siglas en inglés)/EC (siglas en inglés) (un grupo que protege los derechos y el bienestar de las personas en la investigación) del (insertar nombre del sitio), los Institutos Nacionales de la Salud (NIH), otras entidades de regulación locales, de Estados Unidos e internacionales, el personal del estudio, los monitores del estudio, las compañías farmacéuticas que apoyan este estudio y sus representantes. El Certificado de Confidencialidad no impide que usted revele información sobre usted y su participación en el estudio.

Incluso con el Certificado de Confidencialidad, si el personal del estudio se entera de un posible abuso de menores y/o negligencia o riesgo de daño a usted o a otras personas, estamos obligados a decírselo a las autoridades apropiadas.

## O BIEN

Para TODOS los sitios fuera de los Estados Unidos: Se hará todo lo posible para mantener en reserva su información personal. No le podemos garantizar absoluta confidencialidad. Su información personal puede ser revelada si así lo exige la ley. Ninguna publicación de este estudio usará su nombre o lo/la identificará a usted personalmente.

Sus expedientes pueden ser revisados por el ACTG, OHRP (siglas en inglés), FDA, IRB (siglas en inglés)/EC (siglas en inglés) del (inserte el nombre del sitio), los Institutos Nacionales de la Salud (NIH), otras entidades de regulación locales, de Estados Unidos e internacionales, las agencias regulatorias/de salud nacionales, personal del estudio, monitores del estudio, la compañía farmacéutica que apoya este estudio y sus representantes.

Toda la información recopilada sobre usted como parte del estudio se enviará de forma segura al centro de gestión de datos y estadísticas del ACTG en los Estados Unidos para combinarla con la información de otros participantes en el estudio y realizar un análisis estadístico de los resultados del estudio. No se enviará su nombre ni otros identificadores personales. Su sitio de investigación es responsable de enviar su información de acuerdo con las leyes, regulaciones y políticas de su país y sitio de investigación. (No hay nuevos procedimientos en la obtención de los datos)

Una descripción de este ensayo clínico estará disponible en <a href="https://www.ClinicalTrials.gov">https://www.ClinicalTrials.gov</a>, tal como lo requiere la ley en los Estados Unidos. Este sitio de Internet no incluirá información que pueda identificarlo(a) a usted. Como máximo, el sitio de Internet incluirá un resumen de los resultados. Usted puede consultar este sitio de Internet cuando lo desee.

# ¿QUÉ OCURRE SI NO PODEMOS UBICARLO(A) DURANTE EL ESTUDIO?

En el caso de que usted no pueda ser ubicado(a) después de múltiples intentos por contactarnos con usted, el personal del estudio puede intentar contactarse con usted a través de números de teléfono alternativos de familiares, amigos, del coordinador o de conocidos, obtenidos en el tamizaje y actualizados en cada visita. Si usted no puede ser ubicado(a) a través de los contactos alternativos, intentaremos obtener información sobre usted de otras fuentes, tales como miembros de su familia, otros contactos designados o registros clínicos. El propósito de obtener esta información desde el último contacto es determinar si usted ha fallecido y la causa del fallecimiento, y si usted ha tenido alguna enfermedad cardíaca, accidente cerebrovascular o eventos o procedimientos relacionados con una enfermedad vascular.

#### Contacto con Sus Proveedores de Salud

Los sitios pueden modificarlo según los requisitos locales para obtener registros de atención médica: Como se mencionó antes, actualmente no tenemos datos que nos digan si las **PWH** con un riesgo moderado de sufrir enfermedades cardiovasculares según la calculadora de riesgo ASCVD deberían ser tratados con estatinas. Si usted está en este grupo de riesgo moderado, con un puntaje de riesgo de entre 7.5% y 15%, nos gustaría informar a su(s) proveedor(es) de salud sobre los fundamentos del ensayo, pero necesitamos de su permiso para compartir esta información.

Asimismo, con su autorización, para la cual usted debería firmar un permiso, el personal del estudio puede contactar a sus proveedores de salud en relación con cualquier diagnóstico

clínico que usted pueda desarrollar durante el estudio, incluyendo diagnósticos relacionados con el corazón y otros diagnósticos, tales como VIH, o diagnósticos de riñón, hígado o cáncer.

¿Nos autoriza usted a tomar contacto con su(s) proveedor(es) de salud para compartir información respecto a su puntaje de riesgo cardiovascular y los fundamentos del ensayo, para proveerle(s) de información respecto a los diagnósticos clínicos y hacerle saber a su médico(a) que él/ella podría objetar que usted participe en este estudio dado que usted tiene la probabilidad de recibir el placebo en lugar del tratamiento con estatinas?

| SÍ | NO | Iniciales |
|----|----|-----------|
|----|----|-----------|

# ¿CUÁLES SON MIS COSTOS?

No habrá costos para usted por los medicamentos del estudio, las visitas del estudio, los exámenes físicos, las pruebas de laboratorio u otros análisis que requiere el estudio. Usted, su compañía de seguros o su sistema de salud serán responsables por el costo de su atención médica habitual y por los costos de los medicamentos que no suministre el estudio.

Participar en este estudio puede implicar costos adicionales para usted y su compañía de seguros. En algunos casos, es posible que su compañía de seguros no pague estos costos porque usted está participando en un estudio de investigación.

Se le pagará a usted \_\_\_\_\_ en la visita de ingreso, la visita del mes 1 y en las visitas anuales posteriores, por su participación en el estudio. (El equipo recomienda una compensación a los participantes de \$25 en cada visita anual y en la visita de finalización del estudio. A los sitios se les reembolsará el gasto).

# ¿QUÉ SUCEDE SI SUFRO UNA LESIÓN?

Si usted se lesiona como resultado de su participación en este estudio, se le dará tratamiento inmediato para sus lesiones.

Para todos los sitios: los NIH no tienen ningún mecanismo para proveer una compensación directa por lesiones relacionadas con la investigación.

[Sitios: modificar (si es necesario) e insertar alguna de estas dos declaraciones, según corresponda a su sitio. Si a su sitio se le exige que contrate un seguro para ensayos clínicos (CTI, siglas en inglés), esto se debe indicar en el consentimiento informado].

- Este sitio tiene un seguro para ensayos clínicos. Este seguro permitirá al sitio suministrarle a usted una compensación monetaria si sufre un perjuicio como resultado de su participación en este estudio de investigación. O BIEN
- El costo de este tratamiento se le cobrará a usted o a su compañía de seguros. No hay un programa de compensación ya sea a través de esta institución o de los NIH].

Usted no renunciará a ninguno de sus derechos legales al firmar este formulario de consentimiento.

# ¿CUÁLES SON MIS DERECHOS COMO PARTICIPANTE DE LA INVESTIGACIÓN?

Participar en este estudio es totalmente voluntario. Usted puede elegir no participar en este estudio o dejar este estudio en cualquier momento. Su decisión no tendrá ningún impacto sobre su participación en otros estudios dirigidos por NIH y no implicará ninguna penalidad o pérdida de beneficios a los cuales de otra manera tuviese derecho.

Le diremos sobre cualquier nueva información de este u otros estudios que puedan afectar su salud, bienestar o voluntad de permanecer en este estudio. Si usted quiere conocer los resultados del estudio, hágaselo saber al personal del estudio.

## ¿QUÉ HAGO SI TENGO PREGUNTAS O PROBLEMAS?

Para preguntas sobre este estudio o lesiones relacionadas con la investigación, contacte a:

- Nombre del investigador u otro miembro del personal del estudio
- Número de teléfono de la persona nombrada anteriormente

Para preguntas relacionadas con sus derechos como participante de la investigación, contacte a:

• Nombre o cargo de la persona en la Junta Institucional de Revisión (IRB/EC) u otra organización apropiada para el sitio.

• Número de teléfono de la persona nombrada anteriormente.

## PÁGINA DE FIRMAS

Si usted ha leído este formulario de consentimiento (o el mismo le ha sido explicado), todas sus preguntas han sido contestadas y usted acepta participar en este estudio, por favor firme a continuación.

| Nombre del Participante (letra de imprenta) | Firma del Participante y Fecha |
|---|---|
| Representante Legal del Participante (letra de imprenta) (Según corresponda) | Firma del Representante Legal y Fecha |
| Personal del Estudio que Conduce la Discusión del Consentimiento (letra de imprenta) | Firma del Personal del Estudio y Fecha |
| Nombre del Testigo (letra de imprenta) (Según corresponda) | Firma del Testigo y Fecha |

## APÉNDICE IA: ANEXO DEL MODELO DE CONSENTIMIENTO INFORMADO

Ensayo Clínico Aleatorizado para Prevenir Eventos Vasculares en el VIH - (REPRIEVE) (A5332) Versión FINAL 6.0, 16 de mayo de 2022

## TÍTULO CORTO DEL ESTUDIO: REPRIEVE

Se le solicita a usted que firme este anexo de consentimiento porque está participando en un estudio de investigación en \_\_\_\_\_, titulado "Ensayo Clínico Aleatorizado para Prevenir Eventos Vasculares en el VIH - (REPRIEVE) (A5332)."

El propósito de este anexo es incluir información sobre el intercambio de su información genética desidentificada. "Desidentificada" implica que toda la información que le identifique, por ejemplo, su nombre, número de registro clínico y fecha de nacimiento, ha sido eliminada.

La información genética se obtuvo de la muestra de sangre que se extrajo de usted en la visita de ingreso. Usted estuvo de acuerdo en proporcionar esta muestra en el consentimiento original.

A excepción de las actividades descriptas en este anexo, los términos de su formulario de consentimiento original permanecen en plena vigencia, lo que incluye que los resultados del estudio de investigación no les serán entregados a sus familiares, compañías de seguros o empleadores sin su permiso por escrito y la aprobación de la Junta Institucional de Revisión/Comité de Ética en

Por favor, lea atentamente este anexo de consentimiento y tómese su tiempo para tomar una decisión. Cuando el/la médico(a) o el personal del estudio hable con usted de este anexo, pídales que le expliquen cualquier palabra o información que usted no entienda con claridad. No es necesario que firme este anexo para poder permanecer en REPRIEVE (A5332).

## INTERCAMBIO DE SU INFORMACIÓN GENÉTICA

La enfermedad y la salud se ven afectadas por los genes o la información genética que tenemos dentro de nosotros. La información genética que obtenemos en este estudio puede ayudar a avanzar en otros tipos de investigación. Los Institutos Nacionales de la Salud (NIH) han establecido un programa que permite a los investigadores compartir la información genética de diferentes estudios para ayudarnos a conocer más de cada estudio financiado por los NIH. Su información genética se compartirá con otros investigadores a través de una base de datos segura y de acceso controlado respaldada por los NIH.

Cuando compartamos su información genética con otros investigadores a través de una base de datos segura y de acceso controlado respaldada por los NIH, incluidos los estudios del genoma completo (como la determinación de su secuencia de ADN completa en una sola vez), eliminaremos toda la información que le identifique. Esta información desidentificada podrá utilizarse en otras investigaciones. No creemos que

haya más riesgos para su privacidad y confidencialidad al compartir su información genética con esta base de datos de acceso controlado. Sin embargo, no podemos predecir cómo se utilizará la información genética en el futuro.

Su nombre u otra información directamente identificable no se facilitará a la base de datos de acceso controlado respaldada por los NIH. Existen muchas otras salvaguardas para proteger su información mientras se almacena en la base de datos de acceso controlado y se utiliza para la investigación. Aun así, es posible que en el futuro alguien pueda volver a identificar su información. Además, utilizando la base de datos de acceso controlado, los investigadores pueden publicar o presentar los resultados combinados de su investigación, pero no incluirán su nombre ni otra información que pueda identificar a usted.

No se espera que la investigación que utilice su información genética le aporte ningún beneficio directo. Usted puede retirar su consentimiento para compartir su información genética en cualquier momento. Sin embargo, no podemos recuperar ninguna información que ya se haya compartido.

| ¿Acepta compartir su | ı informacióı | n genética? |
|----------------------|---------------|-------------|
| SÍ | NO | Iniciales |

## OTRA INFORMACIÓN

El resto de la información contenida en el consentimiento de REPRIEVE (A5332) que usted firmó también se aplica a este anexo del consentimiento. Se le brindará a usted como referencia una copia firmada de este consentimiento en el momento en que usted brinde su consentimiento a la información de este anexo.

#### PREGUNTAS RESPECTO A ESTE ANEXO DEL CONSENTIMIENTO

Si usted tiene preguntas, preocupaciones o quejas con respecto a este anexo del consentimiento, contacte a el/la Dr. (nombre) al (número) durante el horario de atención al público, y al (localizador) después de hora y en fines de semanas o días festivos.

Para preguntas respecto a sus derechos como participante en la investigación, o para discutir preguntas, preocupaciones o sugerencias relacionadas con la investigación de este anexo del consentimiento, o para obtener información u ofrecer aportes sobre la investigación, contacte a la Junta Institucional de Revisión/Comité de Ética de al (número).

## DECLARACIÓN DE CONSENTIMIENTO

"Se me ha explicado la finalidad de este anexo del consentimiento. Se me ha permitido hacer preguntas, y mis preguntas han sido respondidas a mi satisfacción. Se me ha dicho con quién debo ponerme en contacto si tengo preguntas, para hablar de problemas, preocupaciones o sugerencias relacionadas con la investigación o con este anexo, o para obtener información u ofrecer aportes sobre la investigación. He leído este anexo y acepto las opciones que he indicado anteriormente, entendiendo que puedo retirar mi consentimiento en cualquier momento. Se me ha informado que se me entregará una copia firmada y fechada de este anexo."

## PÁGINA DE FIRMAS

Si ha leído este formulario de consentimiento (o se lo han explicado), si ha respondido a todas sus preguntas y acepta participar en este estudio, firme con su nombre a continuación.

| Nombre del Participante<br>(letra de imprenta) | Firma del Participante y Fecha |
|---|---|
| Representante Legal del Participante<br>(letra de imprenta) (Según corresponda) | Firma del Representante Legal y Fecha |
| Personal del Estudio que Dirige la<br>Discusión del Consentimiento<br>(letra de imprenta) | Firma del Personal del Estudio y Fecha |
| Nombre del Testigo (letra de imprenta) | Firma del Testigo y Fecha |